CLINICAL TRIAL: NCT05699408
Title: A Randomized, Open-Label, Controlled, Parallel-group, Multicenter Trial Comparing the Efficacy and Safety of INS068 and Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled With Oral Antidiabetic Drugs
Brief Title: To Compare the Efficacy and Safety of INS068 and Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled With Oral Antidiabetic Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS068-302
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Controlled, Parallel-group, Multicenter Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INS068 injection (Experimental)
  Interventions: Drug: INS068 injection
- Insulin Glargine (Active Comparator)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: INS068 injection — INS068 injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: INS068 injection
Drug: Insulin Glargine — Insulin Glargine injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: Insulin Glargine

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of INS068 once daily (QD) in subjects with type 2 diabetes not adequately controlled with oral antidiabetic drugs compared to insulin Glargine QD for 26+26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes ≥ 6 months；
2. Stable daily dose(s) for ≥8 weeks prior to screening of any of the following anti-diabetic drug(s) or combination regimen(s): 1) Any metformin formulations ≥1500 mg daily or maximum tolerated (≥1000mg daily). 2) Any of the following oral antidiabetic drugs with dose ≥half of the maximum approved dose according to local label or maximum tolerated): Sulfonylureas, Meglitinides (glinides), dipeptidyl peptidase-4 (DPP-4) inhibitors, Sodium-glucose co-transporter-2 (SGLT2) inhibitors, Thiazolidinediones and Alpha-glucosidase inhibitors.
3. Glycated hemoglobin was 7.0%~11.0% (both inclusive) at screening

Exclusion Criteria:

1. Known or suspected allergy or intolerance to the investigational medicinal products or related products；
2. Hospitalization for diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome during the previous 6 months；
3. Potentially unstable diabetic retinopathy or maculopathy requiring treatment (e.g., laser, surgical treatment or injectable drugs) during the previous 6 months；
4. Have used insulin therapy anytime in the past 2 years, except for short-term insulin treatment and prior treatment for gestational diabetes.
5. Participation in any clinical trial of an approved or non-approved investigational product/treatment within the last 1 month or 5 half-lives, whichever is longer, prior to screening;
6. Women who are pregnant, breastfeeding or planning to conceive, or women of childbearing potential are reluctant to use appropriate contraception during the trial and for at least 14 days after the last dose of the investigational medicinal drug;
7. Any conditions that the Investigator judges might not besuitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 26
  Change from baseline in Glycosylated Haemoglobin after 26 weeks of treatment

SECONDARY OUTCOMES:
Change in FPG(fasting plasma glucose) | Week 0 to Week 26, Week 0 to Week 52
  Change from baseline in FPG after 26 weeks and 52 weeks of treatment
Proportion of Subjects with HbA1c<7% and HbA1c≤6.5% | Week 0 to Week 26 、Week 0 to Week 52
  Proportion of subjects with HbA1c<7% and HbA1c≤6.5% after 26 weeks and 52 weeks of treatment
Proportion of Subjects achieving HbA1c targets (HbA1c<7%; HbA1c≤6.5%) and without grade 2 or 3 hypoglycaemia in the last 12 weeks of the treatment period | Week 0 to Week 26, Week 0 to Week 52
Change in HbA1c | Week 0 to Week 52
per-breakfast SMPG | Week 0 to Week 26 、Week 0 to Week 52
8-point SMPG profiles | Week 0 to Week 26 、Week 0 to Week 52
Average daily Insulin dose | Week 0 to Week 26 、Week 0 to Week 52
Proportion of Subjects requiring rescue therapy during treatment | Week 0 to Week 26 、Week 0 to Week 52
Frequency and severity of adverse events | Week 0 to Week 52 + 14 days follow-up
Incidence and rate of Hypoglycemic events | Week 0 to Week 52 + 14 days follow-up
Change in weight | Week 0 to Week 26、Week 0 to Week 52
Anti-drug Antibodies | Week 0 to Week 52 + 14 days follow-up
Serum INS068 concentration | Week 0 to Week 52
Change in scores of diabetes treatment satisfaction questionnaire status version (DTSQs) | Week 0 to Week 26 、Week 0 to Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided